CLINICAL TRIAL: NCT06316869
Title: Clinical Study of Noninvasive Prediction of Portal Hypertension in Cirrhosis Based on Sound Touch Viscoelastography
Brief Title: Noninvasive Prediction of Portal Hypertension in Cirrhosis Using Sound Touch Viscoelastography
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: STVi
Record Dates: First submitted 2024-03-10; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Portal Hypertension; Cirrhosis
Keywords: Sound Touch Viscoelastography; Clinically Significant Portal Hypertension; Portal Venous Pressure Gradient; Cirrhosis
MeSH Terms: conditions — Hypertension, Portal; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CSPH group: HVPG≥10 mmHg
- Non-CSPH group: HVPG<10 mmHg

SUMMARY:
The objective of this observational study is to investigate and validate the utility of the Sound Touch Viscoelastography(STVi) technique in patients with liver cirrhosis for noninvasive prediction of Portal hypertension (PH). The primary research questions it seeks to address are as follows:

* What is the correlation between the liver STVi index and Portal Venous Pressure Gradient (HVPG)?
* Is STVi an available tool to non-invasively predict PH in patients with liver cirrhosis? And the effectiveness and practicality of STVi will be validated.
* To establish a predictive model for Clinically Significant Portal Hypertension (CSPH) utilizing liver STVi index as the primary indicator.

The HVPG is considered as the gold standard in our study and STVi was employed to quantify the STVi index of the liver in patients with liver cirrhosis. Researchers will compare the two patients groups, HVPG≥10 mmHg and HVPG<10 mmHg, to see the usage of STVi in the noninvasive prediction of PH.

DETAILED DESCRIPTION:
1. Research subjects: Subjects were included in strict accordance with the preparation procedures (inclusion criteria, informed consent), and with the approval of the Ethics Committee of the First Affiliated Hospital of Wenzhou Medical University, relevant data were collected within 1 week after the patients were enrolled and before the HVPG test..
2. Clinical baseline information and laboratory data: including name, gender, age, blood pressure, BMI (height, weight), causes of liver cirrhosis and other general information, and relevant laboratory tests, including platelet count, hemoglobin, albumin, prothrombin time, international normalized ratio, total bilirubin, creatinine, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, blood ammonia, etc.
3. Conventional gray-scale ultrasound and color Doppler examination: including hepatic artery inner diameter, hepatic artery peak flow velocity, hepatic artery resistance index, portal vein trunk inner diameter, portal vein average flow velocity, spleen size, etc.
4. STVi detection: Use the color Doppler ultrasound system (including elastic components) of Shenzhen Mindray Biomedical Electronics Co., Ltd., equipped with an abdominal convex array probe with a probe frequency of 1~6 MHz. The probe was placed in a supine position or slightly tilted to the left, with the right arm raised and fully abducted to increase the width of the intercostal space, and the liver viscoelastic index of the right lobe of the liver was measured between the intercostals. During measurement, the subject should hold his breath for 3 to 5 seconds in a calm state. Do not hold his breath after taking a deep breath. The sampling frame should be placed in a place with uniform echo in the liver parenchyma, avoiding large blood vessels, bile ducts and ribs. The sampling frame should be as parallel to the liver capsule as possible and placed 1 to 2 cm below the liver capsule and no more than 6 cm. The region of interest is preferably placed in the center of the elastogram, and the diameter of the sampling frame is recommended to be ≥1.5 cm. Take the median after 3 valid measurements of the same site. The sampling results require measurement success rate ≥60% and IQR/Median≤0.3.
5. HVPG detection: Use the right jugular vein approach, refer to the Chinese Expert Consensus on Clinical Application of Hepatic Venous Pressure Gradient (2018 Edition) , and select the balloon catheter to the hepatic vein under fluoroscopy, at a distance from the inferior vena cava 2~4 cm, wait at least 20 s (some patients may take longer to reach a stable reading), and then read the Free Hepatic Venous Pressure (FHVP) after the pressure value is stable. After injecting contrast medium or air to expand the balloon to fully block the hepatic venous blood flow, wait at least 40 s until the pressure value is stable, and then read the Hepatic Venous Wedge Pressure (WHVP). Keep the balloon in the inflated state, instruct the patient to hold his breath, slowly inject 5 ml of contrast agent through the balloon catheter, and perform hepatic venography to confirm that there is no contrast agent reflux or venous-venous collateral shunt. Calculated according to the formula HVPG = WHVP - FHVP, HVPG should be the average of 2 measurements.
6. Group according to the HVPG test results and divide them into 2 groups: CSPH group (HVPG≥10 mmHg) and non-CSPH group (HVPG<10 mmHg).
7. Build a model: Screen out independent variable information related to the occurrence of CSPH through model variable screening and correlation analysis, and use it to build a prediction model. And establish a Nomogram model to realize the visualization of the model.
8. Evaluate the model: Discrimination of the model: ROC curve analysis, C-index; Calibration of the model: Hosmer-Lemeshow goodness of fit test, consistency curve (test); Clinical net benefit assessment: Decision curve analysis ( DCA).

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years.
* Clinically diagnosed with cirrhosis. Meeting the diagnostic criteria of the 2019 edition of the "Cirrhosis Diagnosis and Treatment Guidelines": (1) Histology consistent with cirrhosis diagnosis; (2) Endoscopy shows esophageal gastric varices or ectopic varices, excluding non-cirrhotic portal hypertension; (3) Imaging examinations such as ultrasound, LSM, or CT suggest features of cirrhosis or portal hypertension: such as splenomegaly, portal vein ≥1.3 cm, LSM measurements meeting diagnostic thresholds for cirrhosis of different etiologies; (4) In the absence of histology, endoscopy, or imaging examinations, the following abnormal indicators suggest the presence of cirrhosis (must meet 2 of the 4 criteria): a. PLT <100×10^9/L, with no other explanations; b. Serum ALB <35 g/L, excluding malnutrition or other causes such as renal disease; c. INR >1.3 or prolonged PT (discontinuation of thrombolytics or anticoagulants for >7 days); d. AST/PLT ratio index (APRI): Adult APRI score >2, with attention to the influence of hepatotoxic drugs and other factors on APRI.
* Planning to undergo HVPG testing and meeting the indications for HVPG testing in the "Chinese Expert Consensus on the Clinical Application of Hepatic Venous Pressure Gradient (2018 edition)" : (1) Assessing the efficacy of drug therapy for primary and secondary prevention of esophageal gastric variceal bleeding; (2) Predicting the risk of esophageal gastric variceal bleeding and guiding treatment plan selection; (3) Predicting the risk, degree of progression, and clinical prognosis of decompensated events in cirrhosis; (4) Evaluating the efficacy of related new drugs; (5) Evaluating the accuracy of related non-invasive techniques; (6) Diagnosis and differential diagnosis of portal hypertension types.
* Able to understand and voluntarily sign a written informed consent form.

Exclusion Criteria:

* Post-TIPS procedure;
* Post-hepatectomy splenectomy;
* Hepatic malignancy;
* Portal vein thrombosis;
* Individuals with severe cardiac, pulmonary, hepatic, or renal dysfunction;
* Pregnant and postpartum women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Portal Hypertension (PH) is the primary consequence of liver cirrhosis and a crucial factor leading to severe complications such as ascites, rupture and bleeding of esophageal and gastric varices (EGV), and hepatic encephalopathy. It annually results in a significant number of deaths, posing a serious threat to life and health. In China, there is a large population of PH patients, and the long-term follow-up and treatment processes require substantial medical resources. Currently, there is no reliable non-invasive method for convenient and rapid monitoring of portal vein pressure in PH patients. This hinders timely clinical intervention and compromises patient prognosis.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
STVi index | baseline, pre-intervention
  The abdominal convex array probe equipped with the color Doppler ultrasound system (including elastic components) was used to measure the shear wave signals. And then using pulse wave technology and specific computer algorithms (mainly utilizing the Voigt model to calculate liver shear wave viscosity and linear dispersion model to compute shear wave dispersion slope), liver STVi index can be calculated. Since the STVi index is a new evaluation index based on a new ultrasonic technology, there is no clear maximum and minimum values has been reported. Based on previous research, we estimate STVi index was an independent risk factor for high HVPG and was significantly higher in CSPH group than non-CSPH group.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital the First Affiliated Hospital, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No